CLINICAL TRIAL: NCT04268797
Title: Efficacy and Safety of High-frequency Repetitive Transcranial Magnetic Stimulation With H7-coil in the Treatment of Schizophrenia Negative Symptoms; A Multicenter, Randomized, Sham Controlled, Triple Blind Trial
Brief Title: TMS in Treatment of Schizophrenia Negative Symptoms
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sveti Ivan Psychiatric Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TMS_negative symptoms
Record Dates: First submitted 2020-02-07; First posted 2020-02-13 (Actual); Last update posted 2022-05-19 (Actual); Status verified 2022-05

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HR rTMS H7-coil intervention group (Experimental)
  Interventions: Device: HR rTMS
- sham control group (Sham Comparator)
  Interventions: Device: sham

INTERVENTIONS:
Device: HR rTMS — high frequency repetitive transcranial magnetic stimulation (HF rTMS) with H7-coil applied once daily during the twenty days
  Arms: HR rTMS H7-coil intervention group
Device: sham — SHAM HF rTMS coil once daily x 20 days
  Arms: sham control group

SUMMARY:
Primary objective: to examine the efficacy and safety of high frequency repetitive transcranial magnetic stimulation (HF rTMS) with H7-coil applied once daily during the twenty days, augmentative to the standard antipsychotic pharmacotherapy and other treatment of negative symptoms in schizophrenia.

Targeted population: patients diagnosed with schizophrenia, 18-55 years old with predominant negative symptoms, stable condition for >3 months and unchanged antipsychotic therapy for >1 months and no treatment with antidepressants.

Study design: industry independent, multicenter, prospective randomized sham-controlled, two-arms, triple-blind superiority clinical trial with concealed allocation and masked independent outcome assessment.

Primary outcome: adjusted median of differences in total SANS score. Adjustment for age, gender, baseline total SANS score, duration of the disorder, and antipsychotic therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Confirmation diagnosis of schizophrenia (ICD-10 F20) using the Mini-International Neuropsychiatric Interview (MINI) (Lecrubier et al., 1997; Sheehan et al., 1998),
2. Age 18-55 years,
3. Both genders,
4. PANSS negative symptoms subscale score >24,
5. PANSS positive symptoms subscale score <20,
6. Stable condition (no acute psychosis exacerbation, no psychiatric hospitalization because of relapse or worsening of symptoms) during at least three months,
7. Stable antipsychotic therapy with no change of drugs or doses during the one months before the enrollment.

Exclusion Criteria:

1. Antipsychotics dose change or change of antipsychotic drug,
2. Hospitalization for somatic illness in another institution,
3. Termination of treatment in a Psychiatric Hospital "Sveti Ivan",
4. Pregnancy,
5. Missed more than three consecutive interventions,
6. Withdrawal of consent to participate for the sake of intolerance of TMS or for other reasons.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 104 (Estimated)
Dates: Start 2019-11-04 (Actual); Primary Completion 2022-12-15 (Estimated); Study Completion 2023-03-15 (Estimated)

PRIMARY OUTCOMES:
Adjusted median of differences in total SANS score | assessed up to 20 days of treatment
  Adjusted median of differences in total SANS score (Andreasen, 1989). We will adjust the medians for age, gender, baseline total SANS score, duration of the disorder, and antipsychotic therapy

SECONDARY OUTCOMES:
Change in SNS score | assessed up to 20 days of treatment
  Change in Self-Evaluation of Negative Symptoms Scale (SNS) (Dollfus, Mach and Morello, 2016)
Change of BNSS score | assessed up to 20 days of treatment
  Change in Brief Negative Symptom Scale (BNSS), (Kirkpatrick et al., 2006)
Change in PANSS negative symptom subscale with items rescaled to 0-6 range | assessed up to 20 days of treatment
  Change in PANSS negative symptoms subscale with items rescaled to 0-6 range, (Kay, Fiszbein and Opler, 1987)
Change in CDSS score | assessed up to 20 days of treatment
  Change in depressive symptoms measured using Calgary Depression Scale for Schizophrenia (CDSS) (Addington, Addington and Schissel, 1990)

OTHER OUTCOMES:
The number of patients self-reported side effects during therapy, confirmed by the medical nurse | assessed up to 20 days of treatment
Change in verbal memory | assessed up to 20 days of treatment
  Change in verbal memory using Auditory Verbal Learning Test (AVLT), subtest from Wechsler Memory Scale (Revised)-Verbal-Logical Memory
Change in visual memory | assessed up to 20 days of treatment
  Change in visual memory using Benton's visual retention test (BVRT)
Change in numeric memory | assessed up to 20 days of treatment
  Change in numeric memory using subtest from Wechsler Memory Scale (Revised)-Digit Span
Change in visual-spatial abilities and executive function | assessed up to 20 days of treatment
  Change in visual-spatial abilities and executive function using TMT (A/B) Trail Making Test, and subtest from Wechsler Intelligence Scale (Revised)-Block Design
Change in psihomotor speed | assessed up to 20 days of treatment
  Change in psihomotor speed using subtest from Wechsler Intelligence Scale (Revised)-Digit Symbol Substitution Test
Change in verbal fluency | assessed up to 20 days of treatment
  Change in verbal fluency using FAS Verbal Fluency Test
Change in recognition of facial expressions of emotions | assessed up to 20 days of treatment
  Change in recognition of facial expressions of emotions using the Penn's Emotion Recognition Task test (ER40)

CONTACTS AND LOCATIONS:
Locations (1):
- PB Sveti Ivan, Zagreb, Croatia

IPD SHARING:
Plan to Share IPD: No